CLINICAL TRIAL: NCT04076644
Title: Maintenance of Response To Transcranial Magnetic Stimulation (TMS) in Major Depressive Disorder (MDD) Using Monthly TMS Treatment
Brief Title: Maintenance Transcranial Magnetic Stimulation in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Muaid Ithman, Associate Professor of Clinical Psychiatry, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013884
Record Dates: First submitted 2019-08-23; First posted 2019-09-03 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: MDD
Keywords: TMS
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TMS Treatment Arm (Active Comparator): Subjects will receive either a 20min 10hz TMS treatment, or a 3min theta-burst TMS treatment at certain monthly intervals. The TMS treatment protocol they receive depends on what they received in their acute clinical treatment. Subjects in the arm will be tapered off antidepressant medication before TMS treatment begins. Subjects will be assessed monthly for depression using QIDS and PHQ9.
  Interventions: Device: TMS treatment
- No TMS Arm (No Intervention): Subjects will be followed and assessed for depressive symptoms at monthly time intervals similar to the active treatment arm using QIDS and PHQ9. This group does not receive TMS treatment.

INTERVENTIONS:
Device: TMS treatment — TMS using either a standard 10hz 20min or 3 min theta burst protocol
  Other Names: Transcranial Magnetic Stimulation
  Arms: TMS Treatment Arm

SUMMARY:
This an open label study using a FDA-cleared TMS stimulation protocols which will be used to treat patients who have responded or remitted from depression using acute clinical TMS therapy at the University of Missouri-Columbia Neuromodulation Clinic. TMS therapy will be given to subjects at monthly intervals. Depression severity questionnaires will be given monthly to determine if the subjects original response to TMS can be maintained. Subjects will be tapered down from antidepressant medication prior to TMS maintenance treatment. Results will be analyzed to determine the effectiveness and feasibility of maintenance TMS therapies in a clinical setting.

DETAILED DESCRIPTION:
This an open label study using Transcranial Magnetic Stimulation (TMS) as a maintenance treatment for subjects that have seen a clinically significant response or remission from their depressive symptoms after having had an acute clinical course of TMS. All potential subjects must have been treated at the University of Missouri Columbia Neuromodulation Clinic to qualify.

There are 2 arms in this study. The first is a group of patients who will not receive any TMS treatments and will be followed for a year, and have their depression severity assessed monthly using the Personal Health Questionnaire (PHQ9), and the Quick Inventory of Depressive Symptoms.

The second arm will receive TMS treatments 5 times/month for 12 months, be assessed for changes in depressive symptom severity monthly using the PHQ9 and QIDS. TMS treatment protocols will consist of wither the standard 20min 10Hz protocol, or a 3min theta-burst protocol. The protocol used will be determined by what worked for the subject when they were treated clinically at the University of Missouri Columbia Neuromodulation clinic. Subjects in this arm will be tapered of antidepressant medication prior to monthly TMS treatment and will remain antidepressant free for the duration of the study.

The study will be a year long in duration.

ELIGIBILITY:
Inclusion Criteria:

* Must have recently (within 4 weeks) completed an acute TMS course (full 36 treatments) at the University of Missouri Columbia Neuromodulation clinic
* Must have clinically responded to the acute TMS treatment course (≥50% improvement according to the clinical depressive scale used - usually the PHQ-9)
* Must be able sign consent
* Must have a current address and phone number
* Must have current mental health care provider, either psychiatrist or general practioner who they see for mental health symptom management
* Must be able to taper off antidepressant medication before 1st monthly treatment block (treatment group only)

Exclusion Criteria:

* - Subject that has not completed a full acute treatment course, including taper
* Subjects that have changed anything that may not make them safe for TMS, which are (all changes will be reviewed by study MD, and will not necessarily be excluded possibly depending on severity):

  * Any new metal near head
  * Any new medical devices that cannot be removed
  * Any new pregnancies (verbally confirmed)
  * Seizures that occurred post-acute TMS treatment
  * Any uncontrolled cardiovascular disease
  * Any new head trauma
  * Any new illness causing injury to brain
  * Any new medications which cannot be altered or lowered that may be contraindicated for TMS treatment
  * Any drug or alcohol use deemed by the study doctor as unsafe for TMS treatment
* Subjects unwilling to sign consent or follow study procedures
* Subjects with known extended travel plans which may affect study procedures and scheduled TMS treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muaid Ithman, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Neuromodulation Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment were from 8/14/2019 to 5/21/2021. Participants were recruited from outpatient interventional psychiatry clinic at University of Missouri
Pre-assignment Details: Participants had up to 8 weeks to washout of their antidepressant medication, if they could not handle this washout they could not start maintenance treatment. Although two arms were originally planned due to COVID the 2nd arm consisting of group of patients who will not receive any TMS treatments was unable to be recruited.
Period: Overall Study
Arm/Group | TMS Treatment Arm
Started | 11
Completed | 7
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | TMS Treatment Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (16.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity Changes Scored From Patient Health Questionnaire (PHQ9)
Description: The scale was given at the prior to study starting TMS treatments for the study as a baseline measurement. It was then given prior to every monthly TMS treatment block, scale is 0-27 with 0=no depression, 27=severe depression
Time Frame: given at monthly intervals for 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMS Treatment Arm
Number analyzed (Participants) | 7
score on a scale
  Baseline (prior to starting treatment) | 5 (4.04)
  Month 1 | 6.71 (3.05)
  Month 2 | 8.14 (3.18)
  Month 3 | 9.14 (4.67)
  Month 4 | 6.14 (4.22)
  Month 5 | 7.57 (6.06)
  Month 6 | 5.85 (3.09)
  Month 7 | 5.71 (3.49)
  Month 8 | 5.86 (4.26)
  Month 9 | 7.71 (6.12)
  Month 10 | 6.43 (5.12)
  Month 11 | 7.43 (5.83)
  Month 12 | 6.86 (4.55)

2. Primary Outcome: Depression Severity Changes Scored From Quick Inventory of Depression Symptom Questionnaire (QIDS) Pre Treatment Monthly Scores
Description: The scale was given at the prior to study starting TMS treatments for the study as a baseline measurement. It was then given prior to every monthly TMS treatment block (Pre Trt Month) and after every monthly TMS treatment block (Post Trt Month) ,scale is 0-27 with 0=no depression, 27=severe depression
Time Frame: given at baseline and before and after TMS treatment block for 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMS Treatment Arm
Number analyzed (Participants) | 7
score on a scale
  Baseline | 4.14 (2.36)
  Pre Trt Month 1 | 7.57 (3.33)
  Pre Trt Month 2 | 8.86 (4.09)
  Pre Trt Month 3 | 8.43 (4.27)
  Pre Trt Month 4 | 6.86 (4.55)
  Pre Trt Month 5 | 8.86 (5.67)
  Pre Trt Month 6 | 7 (6.07)
  Pre Trt Month 7 | 5.43 (2.82)
  Pre Trt Month 8 | 6.29 (3.41)
  Pre Trt Month 9 | 8.71 (5.90)
  Pre Trt Month 10 | 6.86 (5.17)
  Pre Trt Month 11 | 7.57 (4.66)
  Pre Trt Month 12 | 8.71 (4.91)

3. Primary Outcome: Depression Severity Changes Scored From Quick Inventory of Depression Symptom Questionnaire (QIDS) Post Treatment Monthly Scores
Description: as for outcome 2
Time Frame: given at baseline and before and after each TMS treatment block for 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMS Treatment Arm
Number analyzed (Participants) | 7
score on a scale
  Baseline | 4.14 (2.36)
  Post Trt Month 1 | 6.29 (2.60)
  Post Trt Month 2 | 6 (2.39)
  Post Trt Month 3 | 5.43 (2.44)
  Post Trt Month 4 | 4.55 (4.06)
  Post Trt Month 5 | 6.14 (3.72)
  Post Trt Month 6 | 4.71 (3.88)
  Post Trt Month 7 | 5 (2.53)
  Post Trt Month 8 | 5.43 (3.02)
  Post Trt Month 9 | 6.57 (4.56)
  Post Trt Month 10 | 5 (4.14)
  Post Trt Month 11 | 5.57 (3.42)
  Post Trt Month 12 | 5.43 (3.29)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | TMS Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Due to changes in staff and start of COVID our recruitment was limited. Orginally a non-TMS treatment arm was planned but due to COVID we were unable to recruit for this arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT04076644/Prot_000.pdf